CLINICAL TRIAL: NCT06641297
Title: White Matter Plasticity in Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HP-00081020
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia Disorders
Keywords: music; training; plasticity
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active training (Active Comparator): Training sessions involving playing the video game 'Guitar Hero'
  Interventions: Behavioral: Music video game
- Observation training (Placebo Comparator)
  Interventions: Behavioral: Music video game

INTERVENTIONS:
Behavioral: Music video game — The video game 'Guitar Hero' will be used as the platform for training for participants to acquire a new 'skill'

SUMMARY:
Schizophrenia spectrum disorders are associated with impairment in the microstructure of white matter, the key brain tissue responsible for fast communication between different brain regions necessary for any complex task. This white matter impairment is linked to problems with cognition in schizophrenia, especially slower processing speed. This project aims to study the potential for correcting white matter deficits in schizophrenia by examining mechanisms underlying white matter structure changes in response to training on playing a mock musical instrument.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, or psychosis NOS
* age 15-45
* able to provide informed consent

Exclusion Criteria:

* contraindications to MRI (metal implants, claustrophobia)
* medical condition that limits use of hands (ie, arthritis)
* Active or recent (within 6 months) substance use disorder other than nicotine

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
White matter microstructure | 3 weeks
  fractional anisotropy of white matter tracts as assessed with diffusion tensor imaging

SECONDARY OUTCOMES:
Brain level of N-acetylaspartate | 3 weeks
  NAA levels in motor cortex of brain as measured with magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Maryland Psychiatric Research Center, Catonsville, Maryland
  - University of Maryland Baltimore - Maryland Psychiatric Research Center, Catonsville, Maryland

IPD SHARING:
Plan to Share IPD: No